CLINICAL TRIAL: NCT05842122
Title: Pharmacy Delivery to Expand the Reach of PrEP in Kenya: Cluster-randomized Control Trial
Brief Title: Pharmacy-based PrEP Delivery in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Kenya Medical Research Institute (Other); Jhpiego (Other)
Responsible Party: Principal Investigator, Katrina Ortblad, Assistant Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG1123165; BMGF INV-033052 (Other Grant/Funding Number: Bill & Melinda Gates Foundation); 11136 (Other: Fred Hutchinson Cancer Center IRB)
Record Dates: First submitted 2023-04-05; First posted 2023-05-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hiv
Keywords: Kenya; HIV pre-exposure prophylaxis (PrEP) delivery; PEP; Pharmacy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: In the cluster-randomized control trial, the intervention will be introduced in a parallel fashion (i.e., all pharmacies assigned a given intervention will receive the intervention at the start of the trial).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Client-sustained delivery of pharmacy PrEP/PEP (Active Comparator): Pharmacy providers offer clients PrEP and PEP services for a fee of 250 Kenyan Shillings (KES) per visit (study team compensates pharmacy providers 0 KES per visit).
  Interventions: Behavioral: Client-sustained delivery of pharmacy PrEP/PEP
- Implementor-sustained delivery of pharmacy PrEP/PEP (Active Comparator): Pharmacy providers offer clients PrEP and PEP services for a fee of 0 KES per visit (study team compensates pharmacy providers 250 KES per visit).
  Interventions: Behavioral: Implementor-sustained delivery of pharmacy PrEP/PEP
- Counselor-supported delivery of pharmacy PrEP/PEP (Active Comparator): HIV testing service (HTS) counselors support pharmacy providers in offering clients PrEP and PEP services for a fee of 0 KES per visit (study team compensates pharmacy providers 100 KES per visit).
  Interventions: Behavioral: Counselor-supported delivery of pharmacy PrEP/PEP
- Referral to clinic-based PrEP/PEP (Active Comparator): Pharmacy providers offer clients referral to PrEP and PEP services at nearby public clinics for a fee of 0 KES per referral (study team compensates pharmacy providers 100 KES per referral).
  Interventions: Behavioral: Referral to clinic-based PrEP/PEP

INTERVENTIONS:
Behavioral: Client-sustained delivery of pharmacy PrEP/PEP — * Services delivered: 1) behavioral HIV risk assessment (+ counseling), 2) PrEP/PEP medical safety assessment, 3) HIV testing, and 4) PrEP (30-day supply at initiation; 90-day supply at refill visits) or PEP dispensing (28-day supply) among those determined eligible.
  * Service provider(s): pharmacists or pharmaceutical technologist trained on PrEP/PEP service delivery
  * Cost to client: 250 KES per pharmacy PrEP/PEP visit
  * Payment to pharmacy:* 0 KES per pharmacy PrEP/PEP visit *Pharmacies paid by the research team (i.e., the "implementer" in this trial)
  Arms: Client-sustained delivery of pharmacy PrEP/PEP
Behavioral: Implementor-sustained delivery of pharmacy PrEP/PEP — * Services delivered: 1) behavioral HIV risk assessment (+ counseling), 2) PrEP/PEP medical safety assessment, 3) HIV testing, and 4) PrEP (30-day supply at initiation; 90-day supply at refill visits) or PEP dispensing (28-day supply) among those determined eligible.
  * Service provider(s): pharmacists or pharmaceutical technologist trained on PrEP/PEP service delivery
  * Cost to client: 0 KES per pharmacy PrEP/PEP visit
  * Payment to pharmacy:* 250 KES per pharmacy PrEP/PEP visit *Pharmacies paid by the research team (i.e., the "implementer" in this trial)
  Arms: Implementor-sustained delivery of pharmacy PrEP/PEP
Behavioral: Counselor-supported delivery of pharmacy PrEP/PEP — * Services delivered: 1) behavioral HIV risk assessment (+ counseling), 2) PrEP/PEP medical safety assessment, 3) HIV testing, and 4) PrEP (30-day supply at initiation; 90-day supply at refill visits) or PEP dispensing (28-day supply) among those determined eligible.
  * Service provider(s): pharmacists or pharmaceutical technologist trained on PrEP/PEP service delivery with support from a HTS counselor (to assist with screening and HIV testing)
  * Cost to client: 0 KES per pharmacy PrEP/PEP visit
  * Payment to pharmacy:* 100 KES per pharmacy PrEP/PEP visit *Pharmacies paid by the research team (i.e., the "implementer" in this trial)
  Arms: Counselor-supported delivery of pharmacy PrEP/PEP
Behavioral: Referral to clinic-based PrEP/PEP — * Services delivered: 1) behavioral HIV risk assessment (+ counseling), 2) PrEP/PEP medical safety assessment, 3) referral to clinic-based PrEP/PEP services
  * Service provider(s): pharmacists or pharmaceutical technologist trained on PrEP/PEP service delivery
  * Cost to client: 0 KES per pharmacy PrEP/PEP referral
  * Payment to pharmacy:* 100 KES per pharmacy PrEP/PEP referral *Pharmacies paid by the research team (i.e., the "implementer" in this trial)
  Arms: Referral to clinic-based PrEP/PEP

SUMMARY:
A cluster-randomized control trial (cRCT) testing different cost-sharing models for the delivery of HIV pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP) services at private pharmacies in Kenya. The goal is to assess the effect of different pharmacy-based PrEP/PEP service delivery models on PrEP/PEP initiation and continuation outcomes, compared to pharmacy referral to clinic-based PrEP/PEP services (i.e., what is currently allowed in Kenya at the moment without any changes to policies or guidelines). In the cRCT, 60 pharmacies across Central and Western Kenya will be randomized to one of 4 study arms.

DETAILED DESCRIPTION:
Participating study pharmacies will be 1:1:1:1 randomized to either: 1) client-sustained delivery of pharmacy PrEP/PEP services (clients pay 250 KES/visit; study team compensates pharmacies 0 KES/visit); implementor-sustained delivery of pharmacy PrEP/PEP services (clients pay 0 KES/visit; study team compensates pharmacies 250 KES/visit); 3) Counselor-supported delivery of pharmacy PrEP/PEP services (clients pay 0 KES/visit; study team compensates pharmacies 100 KES/visit); or 4) referral to existing clinic-based PrEP/PEP services (clients pay 0 KES/visit; study team compensates pharmacies 100 KES/visit). The primary cRCT outcomes are PrEP initiation and continuation, assessed 60 days following clients first pharmacy PrEP/PEP visit/referral. We will implement the trial for up to 16 months, or longer, depending on achievement of our primary study objectives.

ELIGIBILITY:
Inclusion Criteria:

Pharmacies

* Registered with the Pharmacy and Poisons Board (PPB)
* Must have at least one full-time licensed pharmacist or pharmaceutical technologist on staff
* Must have a private room where HIV testing and PrEP/PEP counseling can occur
* Must be willing to use a study-specific module within a digital platform (Maisha Meds) to record pharmacy PrEP/PEP dispensing
* Owner must agree to allow a trained research assistant to come to the pharmacy on select days to collect data from a random subset of participants
* Owner must agree to allow providers to participate in a monitored WhatsApp group, optional surveys, and optional in-depth interview
* Owner must agree to allow providers to routinely engage with a technical assistant

Pharmacists/HTS counselors

* ≥ 18 years old
* Licensed pharmacist, licensed pharmaceutical technologist, or NASCOP-certified HTS counselor
* Willing to provide PrEP and PEP services, including HIV testing and associated counseling services
* Completed training on PEP/PrEP service delivery at pharmacies, including certification for rapid diagnostic testing
* Able and willing to provide informed consent
* Complete study training
* Willing to use a study-specific module within a digital platform (Maisha Meds) to document PrEP/PEP services rendered

Clients

* ≥ 16 years old
* Interested in being screened for PrEP or PEP
* Meets all criteria to be eligible for pharmacy-delivered PrEP or PEP on the Prescribing Checklist, including being at risk for HIV and not having any medical conditions that might contraindicate PrEP safety
* Able and willing to provide informed consent

Exclusion Criteria:

Clients

* Unwilling to provide a phone number at which an RA can reach them for completing surveys and communicate important study-related information
* Currently enrolled in any other HIV vaccine or prevention trial
* Have a condition that would preclude provision of informed consent, make study participation unsafe, complicate interpretation of outcome data, or otherwise interfere with achieving study objectives

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5808 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
PrEP initiation | 60 days
  The number of participants at each pharmacy that initiated (i.e., were dispensed) PrEP at the pharmacy or clinic within 60 days of initial pharmacy-based screening.
  Comparisons between intervention arms and the control will rely on self-report from the 60-day client survey, while comparisons between intervention arms will employ pharmacy records.
PrEP continuation | 60 days
  The number of participants at each pharmacy that initiated PrEP at the pharmacy or clinic and returned to the pharmacy or clinic and refilled PrEP within 60 days of initial pharmacy-based screening.
  Comparisons between intervention arms and the control will rely on self-report from the 60-day client survey, while comparisons between intervention arms will employ pharmacy records.

SECONDARY OUTCOMES:
PrEP initiation - 270 days | 270 days
  The number of participants at each pharmacy that initiated (i.e., were dispensed) PrEP at the pharmacy or clinic within 270 days of initial pharmacy-based screening
PrEP continuation - 270 days | 270 days
  The number of participants at each pharmacy that initiated PrEP at the pharmacy or clinic and returned to the pharmacy or clinic and refilled PrEP within 270 days of initial pharmacy-based screening (regardless of any gaps in pill coverage)
PrEP continuation - refilled at least twice 270 days | 60 days
  The number of participants at each pharmacy that initiated PrEP at the pharmacy or clinic and refilled PrEP at least twice within 270 days of initial pharmacy-based screening (regardless of any gaps in pill coverage).
PrEP continuation - any stopping/restarting 270 days | 270 days
  The number of participants at each pharmacy that initiated PrEP at the pharmacy or clinic and refilled PrEP more than 7 days after their expected refill date (i.e., stopping and restarting, also referred to as "PrEP reinitiation") within 270 days of initial pharmacy-based screening.
PrEP adherence | 60 days
  The median adherence score (0-100) among participants at each pharmacy who initiated PrEP at the pharmacy or clinic -using the Wilson et al. scale (2020, AIDS)-as measured at 60 days following initial pharmacy screening.
PEP initiation | 60 days
  The number of participants at each pharmacy that initiated (i.e., were dispensed) PEP ≥1 times at the pharmacy or clinic within 3 days, as measured at 60 days following initial pharmacy screening.
PEP initiation - 270 days | 270 days
  The number of participants at each pharmacy that initiated (i.e., were dispensed) PEP ≥1 times at the pharmacy or clinic within 3 days, as measured at 270 days following initial pharmacy screening.
PEP-to-PrEP transition | 60 days
  The number of participants at each pharmacy that successfully completed PEP (tested negative or self-reported testing negative for HIV between 28 and 45 days after initiating PEP at the pharmacy) and initiated PrEP at the pharmacy or clinic as measured at 60 days following initial pharmacy screening.
PEP-to-PrEP transition - 270 days | 270 days
  The number of participants at each pharmacy that successfully completed PEP (tested negative or self-reported testing negative for HIV between 28 and 45 days after initiating PEP at the pharmacy) and initiated PrEP at the pharmacy or clinic as measured at 270 days following initial pharmacy screening.
PrEP-to-PEP transition | 60 days
  The number of participants at each pharmacy that initiated (i.e. were dispensed) PrEP and subsequently initiated PEP at the pharmacy or clinic within 3 days, as measured at 60 days following initial pharmacy screening.
PrEP-to-PEP transition - 270 days | 270 days
  The number of participants at each pharmacy that initiated (i.e. were dispensed) PrEP and subsequently initiated PEP at the pharmacy or clinic within 3 days, as measured at 270 days following initial pharmacy screening.
PrEP/PEP initiation | 60 days
  The number of participants at each pharmacy that initiated (i.e., were dispensed) either PEP or PrEP at the pharmacy or clinic (within 3 days for PEP clients) as measured at 60 days following initial pharmacy screening.
PrEP/PEP initiation- 270 days | 270 days
  The number of participants at each pharmacy that initiated (i.e., were dispensed) either PEP or PrEP at the pharmacy or clinic (within 3 days for PEP clients) as measured at 270 days following initial pharmacy screening.
PrEP/PEP continuation | 60 days
  The number of participants at each pharmacy that (1) initiated PrEP and refilled PrEP or later were dispensed PEP; or (2) initiated PEP and transitioned to PrEP or later were dispensed PEP again as measured at 60 days of initial pharmacy screening.
PrEP/PEP continuation- 270 days | 270 days
  The number of participants at each pharmacy that (1) initiated PrEP and refilled PrEP or later were dispensed PEP; or (2) initiated PEP and transitioned to PrEP or later were dispensed PEP again as measured at 270 days of initial pharmacy screening.
Recurrent PEP use | 60 days
  The number of participants at each pharmacy that were dispensed PEP ≥2 times as measured at 60 days and 270 days of initial pharmacy screening.
Recurrent PEP use- 270 days | 270 days
  the number of participants at each pharmacy that were dispensed PEP ≥2 times as measured at 270 days of initial pharmacy screening.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Malen, MPH, Study Chair — Fred Hutch Cancer Center; Kendall Harkey, MPH, Study Chair — Fred Hutch Cancer Center
Locations (2):
- Kenya (2):
  - Kenya Medical Research Institute, Kisumu
  - Partners in Health & Research Development, Thika

IPD SHARING:
Plan to Share IPD: No
Deidentified data may be available upon request at the discretion of the study PI (Ortblad).

REFERENCES:
- [Derived] Kareithi T, Roche SD, Meisner A, Omollo V, Ong'wen PA, Harkey K, Kiptinness C, Otieno P, Juma L, Malen RC, Anyona MO, Curran K, Banerjee P, Gichuru E, Asewe M, Yu K, Pintye J, Mugambi ML, Shah PD, Sharma M, Were D, Ngure K, Bukusi EA, Ortblad KF; Pharm PrEP cRCT team. Testing different models of pharmacy-based HIV pre- and post-exposure prophylaxis initiation and management in Kenya: protocol for a cluster-randomized controlled trial. Trials. 2025 Dec 30. doi: 10.1186/s13063-025-09384-7. Online ahead of print. PMID 41466427
- [Derived] Kareithi T, D Roche S, Omollo V, Ong'wen PA, Kiptinness C, Otieno P, Juma L, Malen RC, Harkey K, Anyona MO, Curran K, Banerjee P, Gichuru E, Asewe M, Yu K, Pintye J, Mugambi M, Shah PD, Sharma M, Meisner A, Were D, Ngure K, Bukusi EA, Ortblad KF. Testing different models of pharmacy-based HIV pre- and post-exposure prophylaxis initiation and management in Kenya: protocol for a cluster-randomized controlled trial. Res Sq [Preprint]. 2025 Mar 27:rs.3.rs-5968938. doi: 10.21203/rs.3.rs-5968938/v1. PMID 40195998

DOCUMENTS (1):
  • Informed Consent Form (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT05842122/ICF_000.pdf